CLINICAL TRIAL: NCT06307691
Title: Clinical and Radiographic Evaluation of Immediate Implant Placement Using Osseodensification Versus Traditional Drilling Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Mostafa Ibrahim Omar, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11423
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Implant Complication
Keywords: Implant stability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: patients will be randomly selected into either group using computer generated randomization using (www.randomizer.org). The randomized numbers will be allocated to each site in each patient and will be placed in opaque, sealed and sequentially numbered envelopes. patients will be randomly allocated to test and control groups using randomization schedule.
  Masking/blinding:
  * Participants will be blinded
  * Blinding of the operator will be blinded
  * The outcome assessor will be blinded
  * The biostatistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: conventional drilling (Active Comparator): Atraumatic extraction followed by osteotomy preparation. Osteotomy site will be prepared using conventional drills. Implant placement will follow.
  Interventions: Procedure: Conventional drilling
- Intervention: Osseodensification (Active Comparator): Atraumatic extraction followed by osteotomy preparation. Osteotomy site will be prepared using Densah bur. Implant placement will follow.
  Interventions: Procedure: Osseodensification drilling

INTERVENTIONS:
Procedure: Conventional drilling — Atraumatic extraction, followed by sequential drilling using conventional drills
  Arms: Control: conventional drilling
Procedure: Osseodensification drilling — Atraumatic extraction, followed by osteotomy prepared using densah bur (sequential drilling)
  Arms: Intervention: Osseodensification

SUMMARY:
For the purpose of the study, patients will be divided into two groups, i.e., Group A and Group B. In Group (A), 14 immediate implants will be placed using traditional drilling technique, while in Group (B), 14 immediate implants will be placed using OD drilling technique Osseodensification is a system for implant osteotomy preparation, it compresses the cancellous bone around the revolving drills. It largely improves low bone volume by physically increasing the interlocking between the bone and the implant surface. The Densah burs enhances bone density while generating the least amount of heat.

Traditional oversized drilling is the regular manufacturer recommended technique of drilling. It functions by cutting the bone during osteotomy preparation by sharp fluted drills. The undersizing of the preparation allows the implant to partially compact the bone during insertion.

The objective of the current study is to compare between osseodensification drilling protocol versus traditional undersized drilling protocol in immediate implant placement in anterior maxillary region in terms of implant stability.

DETAILED DESCRIPTION:
Preoperative preparation:

A thorough preoperative assessment of all patients will be carried out including history taking, clinical examination and radiographic examination.

10

● History: Each patient will be interviewed in order to obtain a comprehensive history.

● Clinical examination:

Proper intraoral examination will be done to evaluate the following parameters for the tooth of interest:

1. Restorability of the tooth.
2. Relation to adjacent teeth and the available mesio-distal space.
3. Relation to the opposing teeth and the available interarch space. Intraoral examination will be done for all study participants to ensure compliance with the study inclusion criteria.

Full mouth supragingival debridement will be performed for all participants to ensure gingival health. Oral hygiene An impression will be taken for all study participants to create a study cast on which a radiographic stent will be created to allow standardized parallel technique radiographs to be taken for the patient in the study.

Radiographic examination:

* Periapical radiographs will be done to rule out the presence of any periapical infection and evaluate the presence of caries or periodontal disease in the adjacent teeth.
* Cone Beam Computed Tomography (CBCT) will be taken for each patient to assess:

  1. Bucco-lingual width of bone (measured 1 mm below the alveolar crest).
  2. Mesio-distal width of bone.
  3. Corono-apical height of bone.
  4. Presence of labial undercut, dehiscence or fenestration.
  5. Relation to vital structures as nasal floor and maxillary sinus.
  6. Relation to adjacent teeth.

     B. Surgical Procedure:

  <!-- -->

  1. Local anesthesia in which Septocaine (Articaine hydrochloride 4% with 1:100000 Epinephrine) will be administered via buccal and palatal infiltration prior to any surgical procedure.
  2. In both groups, flapless atraumatic tooth extraction will be performed which includes an intrasulcular incision using a 15c blade, then a periotome will be inserted between the root and the surrounding bone in a wedging action around the root. A small sized straight elevator will be used to luxate the root 11
  3. A Lucas curette will be used to clean the extraction socket of any apical pathology and granulation tissue. 4. A periodontal probe will be used to evaluate the integrity of the bone walls and decide whether the minimum bone height required for implant placement is present. 5. Randomization will be broken at this point to determine which treatment the patient will recieve.

     For Group A: (traditional implant placement) ● A pilot drill will be used to create an osteotomy at the base of the socket and decide implant trajectory. implant diameter will be chosen based on the tooth or its socket apical diameter. ● The surgical motor will be set at a speed of 800-1000 rpm and 1:20 reduction torque.
     * Traditional drills will be used in sequence as per the manufacturer recommended protocol.

     For Group B: (Ossedensification protocol) ● Osteotomy will be prepared using Osseodensification drills in sequence as per the manufacturer recommended protocol. ● The surgical motor will be set at a speed of 800-1000 rpm and 1:20 reduction torque.

  6. Implant placement will finally be done by slowly torquing the implant into the osteotomy, placing the implant in a subcrestal position (1-2mm below crestal bone), with a jumping gap at least 2mm from the buccal bone plate.

  7. A healing collar will be placed over the implant to allow the implant healing to be monitored during the early phase of healing.

C. Postoperative care:

Administration of:

1. Antibiotics (Amoxicillin 500 mg orally four times daily for 5 days).
2. Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily for 3 days then whenever needed).
3. Antiseptic mouth rinse (0.2% Chlorhexidine oral rinse) will be prescribed twice per day for two weeks.

12

Patient self-care instructions:

* Avoid any hard brushing and trauma to the surgical site for two weeks.
* Plaque control will be maintained by chlorohexidine for a month after the surgery.
* After this period, patients will be instructed to continue mechanical tooth cleaning again of the treated sites using a soft toothbrush and roll technique for one month in addition to chlorhexidine twice daily.

D. Postoperative radiographs:

A standardized periapical parallel radiograph will be taken 7 days after implant placement to be analyzed to assess crestal bone level, and after 6 and 9 months after surgery [1].

E. Placement of definitive restoration:

Around 6 months, an implant-level impression coping will be seated on to the implant, and a colored resin will be used to capture the soft tissue emergence profile.

A polyvinyl siloxane (PVS) material will be used to transfer the spatial location of the implant. An implant analog will be placed onto the implant level impression coping, and a gypsum soft tissue hybrid master cast will be created to allow laboratory fabrication of a screw-retained definitive restoration.

A definitive screw-retained zirconia crown will be delivered .

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of extraction of a single, unrestorable tooth in the esthetic zone including maxillary anteriors and premolars
* Age range between 20-60 years old
* An intact buccal plate of bone after extraction
* Medically free patients (Brightman. 1994)
* Cooperative patients willing to follow up for the duration of the study.

Exclusion Criteria:

* Acute infection in the implant site
* Patients incapable of maintaining oral hygiene
* Pregnant and nursing female patients
* Smokers (more than 5 cigarettes per day)
* A habit of bruxism
* Periodontal disease
* Subjects who have a systemic disease which affects bone healing as diabetes
* Use of bone metabolism medicines; (Bisphosphonates) .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Implant stability quotient (ISQ) | 1 week, 2 week, 3 weeks, 4 weeks, 6 weeks, 8 weeks, and 12 weeks postoperatively.
  resonance frequency analysis

SECONDARY OUTCOMES:
Crestal bone level | day of the surgery (baseline), at 3 and 6 months postoperatively)
  Parallel technique periapical radiography

CONTACTS AND LOCATIONS:
Overall Officials: Omar M Ibrahim, Master, Principal Investigator — Cairo University; Omnia K Tawfik, Lecturer, Study Chair — Cairo University; Hany El Nahaas, Professor, Study Director — Cairo Unversity
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Derks J, Hakansson J, Wennstrom JL, Tomasi C, Larsson M, Berglundh T. Effectiveness of implant therapy analyzed in a Swedish population: early and late implant loss. J Dent Res. 2015 Mar;94(3 Suppl):44S-51S. doi: 10.1177/0022034514563077. Epub 2014 Dec 11. PMID 25503901
- [Background] Adell R, Lekholm U, Rockler B, Branemark PI. A 15-year study of osseointegrated implants in the treatment of the edentulous jaw. Int J Oral Surg. 1981 Dec;10(6):387-416. doi: 10.1016/s0300-9785(81)80077-4. PMID 6809663
- [Background] Schwartz-Arad D, Chaushu G. The ways and wherefores of immediate placement of implants into fresh extraction sites: a literature review. J Periodontol. 1997 Oct;68(10):915-23. doi: 10.1902/jop.1997.68.10.915. PMID 9358358
- [Background] Gelb DA. Immediate implant surgery: three-year retrospective evaluation of 50 consecutive cases. Int J Oral Maxillofac Implants. 1993;8(4):388-99. PMID 8270307
- [Background] Agliardi E, Panigatti S, Clerico M, Villa C, Malo P. Immediate rehabilitation of the edentulous jaws with full fixed prostheses supported by four implants: interim results of a single cohort prospective study. Clin Oral Implants Res. 2010 May;21(5):459-65. doi: 10.1111/j.1600-0501.2009.01852.x. Epub 2010 Jan 22. PMID 20105197
- [Background] Schwartz-Arad D, Grossman Y, Chaushu G. The clinical effectiveness of implants placed immediately into fresh extraction sites of molar teeth. J Periodontol. 2000 May;71(5):839-44. doi: 10.1902/jop.2000.71.5.839. PMID 10872969
- [Background] Marquezan M, Osorio A, Sant'Anna E, Souza MM, Maia L. Does bone mineral density influence the primary stability of dental implants? A systematic review. Clin Oral Implants Res. 2012 Jul;23(7):767-74. doi: 10.1111/j.1600-0501.2011.02228.x. Epub 2011 Jun 2. PMID 21635560
- [Background] Farronato D, Manfredini M, Stocchero M, Caccia M, Azzi L, Farronato M. Influence of Bone Quality, Drilling Protocol, Implant Diameter/Length on Primary Stability: An In Vitro Comparative Study on Insertion Torque and Resonance Frequency Analysis. J Oral Implantol. 2020 Jun 1;46(3):182-189. doi: 10.1563/aaid-joi-D-19-00145. PMID 32582919
- [Background] Greenstein G, Cavallaro J. Implant Insertion Torque: Its Role in Achieving Primary Stability of Restorable Dental Implants. Compend Contin Educ Dent. 2017 Feb;38(2):88-95; quiz 96. PMID 28156122
- [Background] Trisi P, Berardini M, Falco A, Podaliri Vulpiani M. New Osseodensification Implant Site Preparation Method to Increase Bone Density in Low-Density Bone: In Vivo Evaluation in Sheep. Implant Dent. 2016 Feb;25(1):24-31. doi: 10.1097/ID.0000000000000358. PMID 26584202
- [Background] Boustany CM, Reed H, Cunningham G, Richards M, Kanawati A. Effect of a modified stepped osteotomy on the primary stability of dental implants in low-density bone: a cadaver study. Int J Oral Maxillofac Implants. 2015 Jan-Feb;30(1):48-55. doi: 10.11607/jomi.3720. PMID 25615915
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329